CLINICAL TRIAL: NCT00802217
Title: A Phase 1 Open-Label, Single-Dose, Dose Escalation Study in Healthy Subjects to Evaluate the Safety and Pharmacokinetics of Orally Administered Civamide (Zucapsaicin)
Brief Title: Oral Civamide Safety, Tolerability First in Human Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PK results demonstrated no systemic absorption
Sponsor: Winston Laboratories (Industry)
Responsible Party: Scott B. Phillips, M.D., Winston Laboratories, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WL-1001-03-01
Record Dates: First submitted 2008-11-26; First posted 2008-12-04 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety; Tolerability; Healthy Volunteers
MeSH Terms: interventions — zucapsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Civamide liquid filled softgel capsule 5 mg
  Interventions: Drug: Civamide
- Cohort 2 (Active Comparator): Civamide liquid filled soft gel capsules 2 x 5 mg
  Interventions: Drug: Civamide

INTERVENTIONS:
Drug: Civamide — 5 mg liquid filled softgel capsules
  Other Names: oral civamide
  Arms: Cohort 1
Drug: Civamide — 5 mg x 2 liquid softgel capsules
  Other Names: oral civamide
  Arms: Cohort 2

SUMMARY:
Safety and pharmacokinetic first-time-in-human study of orally administered civamide in healthy subjects.

DETAILED DESCRIPTION:
This is an open-label, non-randomized pharmacokinetic study of two dosage strengths of oral Civamide. The study consists of a Screening Period (Days -21 to Day -2), an Admittance Period, A 4 Day in-house Treatment Period(Days 1-4))and a follow-up Visit on Day 7.

Pharmacokinetics will be assessed at specified timepoints relative to dosing on Day 1 during the in-house stay. Subjects will be discharged from the research unit following the 72 hr blood draw.

Subjects will return to the research unit on Day 7 for a follow-up safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to performing any of the screening procedures.
2. Healthy, determined by pre-study medical evaluation (medical history and physical examination, vital signs, ECG, and clinical laboratory evaluations).
3. Males or females between 18 to 45 years of age, inclusive.
4. Female subjects must be of nonchildbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year) with follicle stimulating hormone [FSH] > 40 U/L).
5. Non-smokers (or other nicotine use) as determined by history (no nicotine use over the past year) and by urine cotinine concentration (< 200 ng/ml) at screening and/or Day -1.
6. Body mass index (BMI) between 18.5 and 30.5 kg/m2, inclusive, at screening.
7. Subject is willing and able to cooperate to the extent required by the protocol.

Exclusion Criteria:

1. Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the Investigator or designee.
2. Subjects with a history or clinical findings of coronary artery disease/cardiovascular disease or ECG findings judged clinically significant by the Investigator.
3. Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
4. Subjects with active upper gastrointestinal problems such as gastroesophageal reflux disease (GERD), or peptic ulcer disease.
5. Subject has known allergy or hypersensitivity to capsicum, Civamide, or capsaicin-containing products.
6. Positive screening test for Hepatitis B surface antigen, Hepatitis C antibody, or HIV antibody.
7. Subject has history of alcohol and/or illicit drug abuse within two years of entry.
8. Positive blood test for ethanol at screening or Day -1.
9. Positive urine drug test (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, tetrahydrocannabinol [THC], etc.) at screening or Day -1.
10. Female subjects of childbearing potential or who are pregnant or breastfeeding.
11. Inability to refrain from consumption of coffee and caffeine containing beverages within 24 hours prior to Day -1 until discharge from the unit on Day 4.
12. Inability to refrain from use of alcohol or alcohol-containing foods, medications or beverages within 48 hours prior to Day -1 until discharge from the unit on Day 4.
13. Topical use of any capsaicin-containing product for 60 days prior to Day -1 until end of study participation.
14. Ingestion of any capsaicin-containing foods (capsicum, cayenne pepper, red pepper, green pepper, Scotch Bonnet, Habanero peppers, African chilies, Tabasco peppers, paprika, pimiento, Mexican chilies, Louisiana long pepper, Louisiana short pepper, Bird pepper, Garden pepper, Goat's pod, Grains of Paradise, Hot pepper, Hungarian Pepper, Ici Fructus, Sweet pepper, and Zanzibar pepper) for 48 hours before Day -1 until end of study participation.
15. Donation of blood (> 250 ml) or blood products within 2 months (56 days) prior to Day -1.
16. Consumption of grapefruit containing food/beverages or Seville oranges (orange marmalade) from 7 days prior to Day -1 until discharge from the unit on Day 4.
17. Use of over the counter (OTC) medications (including vitamins), prescription medications, or herbal remedies from the 14 days prior to Day -1 until discharge from the unit on Day 4. By exception, acetaminophen £ 1 gram per day is permitted and hormone replacement therapy is permitted.
18. Use of an investigational drug within 30 days prior to Day -1.
19. Unwilling to abstain from vigorous exercise from 48 hours prior to Day -1 until discharge from the unit on Day 4.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Measure the absorption of serum Civamide through pharmacokinetics assessments | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Phillips, M D, Study Director — Winston Laboratories; Shwe Gyaw, M D, Principal Investigator — Parexel
Locations (1):
- Parexel International, Inc., Baltimore, Maryland, United States